CLINICAL TRIAL: NCT05594641
Title: Lactate Clearance After Remote Ischaemic Preconditioning in Liver Resections
Brief Title: Lactate Clearance After RIPC in Liver Resection
Acronym: ARAGON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5033
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-11

CONDITIONS: Liver Surgery; Remote Ischaemic Preconditioning
Keywords: lactate clearance; postoperative recovery

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T (Treatment) (Experimental): Remote ischaemic preconditioning (RIPC) will be performed before the start of liver resection and the associated Pringle maneuver
  Interventions: Other: Remote ischaemic preconditioning
- C (Control) (Other): RIPC will be not performed
  Interventions: Other: Control

INTERVENTIONS:
Other: Remote ischaemic preconditioning — A tourniquet will be applied to the right arm and it will be inflated (3 cycles, each lasting 5 minutes, at a pressure of 200 mmHg); each cycle is followed by 5 minutes of resting
  Other Names: RIPC
  Arms: T (Treatment)
Other: Control — The tourniquet will be applied to the right arm but the cuff will be not inflated
  Arms: C (Control)

SUMMARY:
The primary aim of the study is the evaluation of the efficacy of remote ischemic preconditioning (RIPC) in terms of increase of the clearance of lactates 4 hours after the end of the hepatic resection. The secondary aims of the study are represented by the evaluation of the patients' postoperative recovery and the restoration of a normal lactate metabolism.

DETAILED DESCRIPTION:
Hepatic surgery includes clamping of the hepatic peduncle (Pringle maneuver) to control intraoperative bleeding with a consequent reduction of postoperative complications. Surgical manipulations and Pringle maneuver, especially if prolonged and/or repeated, can cause ischemia-reperfusion damage. The technique of regional ischemic preconditioning was introduced to improve tolerance to ischemia. However, the scientific evidence currently does not support the routine use of regional ischemic preconditioning in hepatic surgery. It has recently been demonstrated that ischemic preconditioning can be effective when performed in the upper limb (RIPC). The main advantages of the remote ischaemic preconditiong compared to the regional one are the ease of use, the reduction of surgical time and hepatic ischemia.

One of the most relevant epiphenomena of hepatic ischemia during hepatectomy is an increase in lactate levels in the immediate postoperative period that can be associated with an unfavorable outcome and can affect relevant clinical choices such as admission to intensive care. However, no previous studies have investigated the effectiveness of RIPC in improving lactate clearance after liver resection.

The investigators hypothesized that applying RIPC before the start of the hepatic resection and the associated Pringle maneuvers could significantly increase lactate clearance 4 hours after the end of liver resection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Elective liver surgey (laparotomic, laparoscopic and robotic-assisted)
* Signed informed consent

Exclusion Criteria:

* Age <18 years
* Previous liver intervention including surgical and non surgical approach such as liver radiofrequency ablation and radiation therapy
* Severe cardiopulmunary diseases
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Lactate clearance | 4 hours after the end of liver resection
  (lactate at the end of liver resection minus lactate at 4 hours after the end of liver resection)*100 to lactate at the end of liver resection

SECONDARY OUTCOMES:
Postoperative recovery | hours (RR) or days (ICU), and average of three hours for RR and one day in ICU
  Lenght of stay on recovery room (RR) or in intensive care (ICU)
In-hospital stay | Days until discharge, an average of 7 days
  Hospital stay duration
Trend of lactate clearance | 1, 4 and 24 hours after the end of liver resection
  Repeated measure for lactate clearance

CONTACTS AND LOCATIONS:
Overall Officials: Paola Aceto, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- UOC Anestesia delle Chirurgie Generali e dei Trapianti, Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy